CLINICAL TRIAL: NCT05777408
Title: Additional Effect of Cranial Base Release on Cervical Range and Proprioception in Patients With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/3
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain
Keywords: Range of Motion, Proprioception
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive conventional physical therapy along with Natural apophyseal glides and the second will receive Natural Apophyseal Glides in addition to cranial base release with conventional physical therapy. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants of this group will receive the conventional physical therapy protocol mentioned above. In addition to this, they will receive Natural apophyseal glides 3 sets of 10 repetitions.
  * Frequency: 3 times a week for 2 weeks. 6 sessions in total.
  * Mobilizations will be performed in Grade 1 initially and then progressed to Grade 2 and 3 depending on the patients pain status and compliance.
  Interventions: Procedure: Conventional Physical Therapy; Procedure: Natural Apophyseal glides
- Experimental Group (Experimental): * Participants of this Group will receive the conventional physical therapy protocol mentioned above. In addition to this, they will receive Natural apophyseal glides and cranial base release.
  * Frequency: 3 times a week for 2 weeks. 6 sessions in total.
  * Cranial base release would be given for around 1-4minutes until the tissues relax and would be given once daily
  Interventions: Procedure: Conventional Physical Therapy; Procedure: Natural Apophyseal glides; Procedure: Cranial Base Release

INTERVENTIONS:
Procedure: Conventional Physical Therapy — * 15 mins of TENS (frequency 100 Hz, phase duration 50 μs) with moist heat over the area of pain
  * Isomeric Stretching of neck muscles followed by neck isometrics
Procedure: Natural Apophyseal glides — -Will be applied in sitting position Therapist right hand would cradle the head such that the little finger would rest on the spinous process of the vertebra that is to be mobilized. The other hands thumb would be used to apply over pressure. Direction of force will be parallel to highly irritable-grossly restricted cervical facet joints. Intervention would involve 3 sets of 20 repetitions in 15minutes, 3 days a week for 2 weeks comprising of total 6 session.
Procedure: Cranial Base Release — Will be performed in lying position. therapist fingers will contact the sub occipital muscles and upward pressure would be given until the tissues and muscles relax. it will be given once daily for 3 days a week and will continue for 2 weeks
  Arms: Experimental Group

SUMMARY:
Mechanical Neck pain is the second most commonly occurring musculoskeletal disorder worldwide, ranking 4th in overall disability. It is referred to as Nonspecific generalized neck pain with mechanical characteristics with a primary location between the supranuchal line and the first thoracic spinous process, includingpatients suffering from mechanical neck pain are reported to have several impairments, including pain, reduced cervical ROM, neck disability, and proprioceptive dysfunction. The treatment indicated involves the use of electrotherapy and thermal modalities. In addition, the use of different manual therapy techniques is advocated; however, the most effective management is still debatable. Evidence suggests that Natural Apophyseal glides have a significant positive effect on mechanical neck pain patients. So the study will identify the additional effect of cranial base release with natural apophyseal glides in alleviating pain and its effects on proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mechanical neck pain having reproducible non-specific neck pain with a primary location between the supranuchal line and the first thoracic spinous process
* Male and Female
* Age 18-40 years
* Pain severity on NPRS >3
* Neck Disability score of 20% or above
* Problem not older than 2 months

Exclusion Criteria:

* Patients with history of
* Recent significant trauma (including whiplash)
* Radiculopathy
* Cervical fracture
* Neck surgery
* Dizziness, vertigo
* Myelopathy, Malignancy
* Metabolic disease
* Diagnosed Osteoporosis, Rheumatoid arthritis
* Long-term corticosteroid and/or painkiller drug use

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain | 2 weeks
  Pain will be measured on Numeric Pain Rating Scale.
Change in ROM | 2 weeks
  Cervical rotation will be measured through CROM device
Change in Cervical Proprioception | 2 weeks
  Will be measured from Laser Pointer Method

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan